CLINICAL TRIAL: NCT00722618
Title: Improving Communication With IVF Patients About Risks Such as Multiple Births
Brief Title: Communication With in Vitro Fertilization (IVF) Patients About Risks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 220060957; 1R21HD053459-01A1 (NIH)
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Infertility
Keywords: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Written materials, telephone based education
  Interventions: Behavioral: Written materials, telephone based education
- Comparison (Other): Written materials
  Interventions: Other: Written materials

INTERVENTIONS:
Behavioral: Written materials, telephone based education — 4 new written materials, 15-20 minute educational session by telephone
  Arms: Intervention
Other: Written materials — 2 written materials available on public website
  Arms: Comparison

SUMMARY:
The primary objective of this trial is to determine whether written educational materials plus brief education by telephone will help patients better understand and participate in the decision on how many embryos to transfer to the uterus during treatment of infertility with in vitro fertilization (IVF). The main study hypothesis is that women and men who receive the study's educational intervention will experience favorable changes in knowledge and beliefs about benefits, susceptibility and severity of multiple gestation that impact decisions about the number of embryos to transfer. Secondary objectives are to understand patient beliefs, knowledge and information preferences regarding other possible risks of IVF, to compare perception of IVF-related risks to familiar risks that are included in routine preconception health promotion, and during IVF, and to prepare couples to manage IVF-related obstetrical risks when they make the transition to prenatal care after becoming pregnant.

Medical Treatment Coverage: None, this study does not provide any monetary contribution to medical treatment

DETAILED DESCRIPTION:
The long-term objective of this research is to improve patient understanding of the known and strongly suspected risks from treating infertility with assisted reproductive technologies such as in vitro fertilization (IVF). During IVF, when more embryos are transferred to the uterus, the risk of pregnancy with multiple fetuses increases. In addition, single infants conceived with IVF are at greater risk for low birth weight. This study will promote behaviors that may reduce these risks. One in 3 women who completes a pregnancy conceived with assisted reproductive technologies such as IVF delivers multiples, and these treatments produce over 12,000 multiple birth deliveries annually in the United States. This study will lead to a better understanding of the most effective ways to counsel IVF patients about the embryo transfer decision. This study will also help define how to prepare IVF patients to work most effectively with their prenatal care team to manage IVF-related obstetrical risks.

Medical Treatment Coverage: None, this study does not provide any monetary contribution to medical treatment

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age

Exclusion Criteria:

* Using a gestational carrier in the current cycle of IVF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2007-09; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
questionnaire assessing knowledge, risk perception, self efficacy and preferences, interview about risk perception and decision making | Prior to IVF treatment cycle, 8 weeks

SECONDARY OUTCOMES:
Adoption of healthy preconception behavior, self-efficacy for addressing IVF related obstetrical factors | Prior to IVF treatment cycle, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Linda Frazier, MD, Principal Investigator — University of Kansas School of Medicine-Wichita
Locations (1):
- University of Kansas School of Medicine, Wichita, Kansas, United States